CLINICAL TRIAL: NCT04893057
Title: SARS-CoV-2 sERoprévalences Dans la Population Des Femmes Enceintes et Donneurs de Sang
Brief Title: COVID-19 Seroprevalence in Pregnant Women and Blood Donors
Acronym: CoVERED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/601
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: Women admitted to hospital for a live birth.
- Blood donors: Subjects qualified for whole blood donation

SUMMARY:
The study aims to measure the SARS-CoV-2 seroprevalence (ie. the proportion of people with antibodies against the virus) in pregnant women and blood donors in an administrative area of France, and to determine whether these measures are representative of the general population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

  * Adult female
  * Admitted to hospital for live birth
  * Informed consent
  * Affiliated to the French social security health insurance scheme
* Blood donors

  * Adult male or female
  * Qualified for whole blood donation (up to 70 years old in France)
  * Informed consent
  * Affiliated to the French social security health insurance scheme

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subject without health insurance coverage
* Exclusion period of another study or exclusion period of the French national healthy volunteer registry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult pregnant women and adult blood donors
Sampling Method: Non-Probability Sample
Enrollment: 797 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 spike protein total IgG | at inclusion
  Total IgG directed against anti-SARS-CoV-2 spike protein as measured by ELISA assay

SECONDARY OUTCOMES:
Anti-SARS-CoV-2 nucleocapsid protein total IgG | at inclusion
  Total IgG directed against anti-SARS-CoV-2 nucleocapsid protein as measured by ELISA assay

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Desmarets, MD, PhD, Principal Investigator — CHU Besançon
Locations (1):
- CHU de besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No